CLINICAL TRIAL: NCT04913259
Title: Remote Monitoring for Ambulatory Care of Elderly Patients With Cancer: The TS-PAC Study
Brief Title: Remote Monitoring for Ambulatory Care of Elderly Patients With Cancer
Acronym: TS-PAC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IB 2020-03; 2020-A02584-35 (Other: ANSM IDRCB number)
Record Dates: First submitted 2021-05-20; First posted 2021-06-04 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Cancer
Keywords: Remote monitoring; Elderly patients; Cancer; Ambulatory care
MeSH Terms: conditions — Neoplasms | interventions — Remote Patient Monitoring

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote monitoring for elderly patients with cancer (Other)
  Interventions: Other: Remote monitoring

INTERVENTIONS:
Other: Remote monitoring — Online remote monitoring tool during the care of patients over the age of 65 who are receiving medical treatment for cancer

SUMMARY:
Monocentric, prospective cohort pilot study evaluating the feasibility of a online remote monitoring tool during the care of patients over 65 years of age being medically treated for cancer.

DETAILED DESCRIPTION:
Each patient will have to answer the remote monitoring questionnaires on a mobile phone, tablet or computer via the Internet. Responses will be sent to the referring oncologist and team (Coordinating Nurse). For each question, predetermined response thresholds have been established, triggering "orange" (to watch) or "red" alerts (intervention by the healthcare team required).

In parallel, patient will continue standard follow-up with their referring oncologist and, if necessary (age ≥ 70 years and G8 score ≤ 14), will benefit from an onco-geriatric evaluation at inclusion then at 3 and 6 months.

At the end of 6 months of remote monitoring, the Coordinating Nurse will inform the patient of the end of study participation. Within one month of the end of the remote monitoring, the nurse will also remove the installation of the application and will organize the return of the equipment (tablet and/or 4G LTE key (4th Generation Long Term Evaluation)) if these were lent for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 65 years of age and over.
2. Histologically proven cancer: breast, lung, ovary, prostate, bladder, kidney, ear-nose-throat, colon-rectum, melanoma, sarcoma, lymphoma, myeloma, or myelodysplastic syndrome.
3. Included before starting medical treatment (chemotherapy, hormone therapy, targeted therapy, immunotherapy or combination).
4. Informed consent dated and signed.
5. Patients affiliated with a French social security scheme in accordance with the French law on biomedical research (Article 1121-11 of the French Code of Public Health).

Exclusion Criteria:

Life expectancy less than 12 months. 2. Patient declining to use a tablet, computer, mobile phone or the Internet. 3. Patient not knowing how to read and understand French. 4. Technical impossibility of connecting to the Internet in the patient's living area.

5. Patient already included in this study or in another study evaluating a remote monitoring system.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who completed at least all of 9 questionnaires at 3 months | 3 months

SECONDARY OUTCOMES:
Number of toxicities and clinical symptoms reported by patients triggering a "red" alert. | Weekly during 6 months
  Toxicities and symptoms will be assessed weekly using 20 questions selected and adapted from the French version of the CTCAE PRO (Basch et al., 2014; National Cancer Institute, 2017). For each question, predetermined response thresholds have been established, triggering "orange" (to watch) or "red" alerts (intervention by the healthcare team required). The number of red alerts will be collected for each patient.
Rate of patients according to the compliant score. | Monthly during 6 months
  Patient compliance with oral treatment will be assessed on a monthly basis during the treatment from the self-questionnaire MMAS-4 (Morisky et al., 1986) which has a range from 0 to 4. A high compliant score is defined by a score of 0, a medium compliance score (score=1 or 2) and a low compliance score (score=3 or 4).
Rate of patients with perceived benefit of treatment. | 3 months and 6 months
  The subjective evaluation of the perceived benefit of treatment will be evaluated at 3 and 6 months by a questionnaire developed specifically for this project. It comprises 3 items.The proportion of patients will be reported for each item of the questionnaire.
Rate of patients with satisfaction with the use of the remote monitoring tool | 3 months and 6 months
  Patient satisfaction with the use of the remote monitoring tool will be evaluated at 3 and 6 months by a questionnaire developed specifically for this project. It comprises 2 items. The rate will be reported for each item.
Number of unscheduled hospitalizations> 24 hours and emergency room visits | 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde CABART, Dr, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonie, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No